CLINICAL TRIAL: NCT00781170
Title: Dose-Reduced Allogeneic Stem Cell Transplantation as Induction of a Graft-Versus-Myeloma-Effect After Autologous High-Dose Chemotherapy in Patients With Multiple Myeloma Stage II/III
Brief Title: Dose-Reduced Allogeneic Stem Cell Transplantation After Autologous High-Dose Chemotherapy in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Prof. Dr. N. Kroeger, University Medical Center Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Auto/Allo Plasmozytom
Record Dates: First submitted 2008-10-22; First posted 2008-10-28 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Multiple Myeloma; Stem Cell Transplantation
Keywords: Multiple Myeloma; Plasmocytoma; Stem Cell Transplantation
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: allogeneic hematopoietic SCT

SUMMARY:
To evaluate the feasibility and efficacy of a autologous stem cell transplantation followed by a Melphalan/ Fludarabine based dose-reduced allograft from HLA-identical and HLA-compatible unrelated donor in patients with Multiple Myeloma. In those with non complete remission DLI and/ or new agents such as Bortezomib, Thalidomid or Lenalidomide can be used to upgrade remission.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma Stadium II / III acc. to Salmon and Durie
* signed informed consent
* adequate organ function prior autologous respectively allogeneic SCT
* availability of HLA-identical related or unrelated donor
* availability of at least 2 x 10^6 CD34+ cells per kg BW of recipient for the autologous SCT and at least 3 x 10^6 CD34+ cells for allogeneic SCT
* for MRD-SCT: 18-66 years; for MUD-SCT: 18-55 years
* at age <55 years existence of risk factors that make an myeloablative allogeneic transplantation to risky
* consent of donor to give DLI

Exclusion Criteria:

* severe heart insufficiency
* cardiovascular diseases or severe concomitant diseases
* active infections that need antibiotic therapy
* positive for HIV or hepatitis
* malign secondary disease
* limited liver function with total bilirubin > 1.5 ULN
* increased transaminase > 3 ULN
* increased serum creatinine > 2 mg/dl
* pregnant or lactating women
* known hypersensitivity to Fludarabine or Melphalan
* participation in another trial

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2000-05

PRIMARY OUTCOMES:
Safety and efficacy of a conditioning regimen with Fludarabine, Melphalan and ATG prior allogeneic SCT after high dose chemotheraoie and autologous SCT. Evaluation of underlying disease and donor-recipient-chimerism.

SECONDARY OUTCOMES:
Evaluation of engraftment of leucocytes and platelets
Evaluation of incidence of acute and chronic GvHD
Evaluation of infectious complications
Evaluation of the effects of DLI in case of no CR
Evaluation of disease-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Germany

REFERENCES:
- [Derived] Kroger N, Badbaran A, Zabelina T, Ayuk F, Wolschke C, Alchalby H, Klyuchnikov E, Atanackovic D, Schilling G, Hansen T, Schwarz S, Heinzelmann M, Zeschke S, Bacher U, Stubig T, Fehse B, Zander AR. Impact of high-risk cytogenetics and achievement of molecular remission on long-term freedom from disease after autologous-allogeneic tandem transplantation in patients with multiple myeloma. Biol Blood Marrow Transplant. 2013 Mar;19(3):398-404. doi: 10.1016/j.bbmt.2012.10.008. Epub 2012 Oct 16. PMID 23078786